CLINICAL TRIAL: NCT02845609
Title: A Phase 2 Study to Evaluate the Efficacy of Sialic Acid-Extended Release (SA-ER) Tablets in Patients With GNE Related Thrombocytopenia
Brief Title: Efficacy of Sialic Acid GNE Related Thrombocytopenia
Acronym: SA-thrombo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA thrombo-HMO-CLIT
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2016-07

CONDITIONS: Thrombocytopenia
Keywords: Congenital macrothrombocytopenia; Sialic acid; Bleeding
MeSH Terms: conditions — Thrombocytopenia; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Sialic acid-Extended release 2000 mg, three times per day (TID) for 3 months
  Interventions: Drug: Sialic Acid-Extended Release

INTERVENTIONS:
Drug: Sialic Acid-Extended Release — Oral drug of Sialic acid
  Other Names: aceneuramic acid, UX001

SUMMARY:
Sialic Acid-Extended Release (SA-ER, aceneuramic acid, UX001) is an extended release formulation of sialic acid (SA, also known as N-acetylneuraminic acid or NANA). The SA-ER is currently studied as a substrate replacement therapy for patients with GNE myopathy. The investigators plan to study the SA-ER compound in a cohort of five patients with GNE-related thrombocytopenia.

DETAILED DESCRIPTION:
The investigators identified 5 affected individuals (3 males and 2 females from three families, age 19-40 years) with GNE-related thrombocytopenia . All subjects will receive 2 gram SA-ER, three times per day for a total daily dose of 6 grams (6,000 mg). The dose should be administered with food (i.e. within 30 minutes of a meal or snack).

Efficacy will be evaluated by improvement in clinical and laboratory assessments. Results from Baseline assessments will be compared with those of post-treatment assessments with efficacy conclusions based on improvement between Baseline and the last scheduled assessment. Safety will be evaluated by the incidence and frequency of adverse events, including clinically significant changes from Baseline to scheduled time points in:

* Vital signs.
* History and physical examination findings.
* Laboratory evaluations.
* Serum uric acid levels and urinary excretion of uric acid.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GNE-related macrothrombocytopenia in the investigated family

Exclusion Criteria:

* non consenting for this study
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Increase in platelet count from baseline | 3 month

SECONDARY OUTCOMES:
Incidence and frequency of AEs and SAEs (Safety) | 3 months

IPD SHARING:
Plan to Share IPD: Undecided